CLINICAL TRIAL: NCT03023540
Title: International, Multi-center, Open Label, Follow-up Extension Study Assessing the Long-term Safety and Tolerability of PXT3003 in Patients With Charcot-Marie-Tooth Disease Type 1A
Brief Title: Assessing Long Term Safety and Tolerability of PXT3003 in Patients With Charcot-Marie-Tooth Disease Type 1A
Acronym: PLEO-CMT-FU
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pharnext S.C.A. (Other)
Collaborators: Synteract HCR (Syneos Health) (Unknown); Premier Research (Other); Greenphire (Unknown); Theradis (Unknown); Amarex (Unknown); Eurofins Optimed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLN-PXT3003-03; 2015-002379-81 (EudraCT Number)
Record Dates: First submitted 2016-12-26; First posted 2017-01-18 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Charcot-Marie-Tooth Disease, Type IA
Keywords: Charcot Marie Tooth Type 1A; Peripheral neuropathy; PXT3003
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Patients who completed the pivotal phase III study CLN-PXT3003-02 are allowed to continue in this open-label study. In Period 1, patients who were randomly assigned to placebo or low-dose PXT3003 in pivotal phase III study were assigned to receive low-dose PXT3003 (5 mL), whereas patients assigned to high-dose PXT3003 continued on that dose (receiving the high-dose PXT3003 (5 mL) or twice the low-dose for each administration (i.e. 10 mL)). The primary objective was to assess safety and tolerability for prolonged exposure to PXT3003, and to evaluate the effect on disability in patients with mild to moderate CMT1A.
  In Period 2, all patients are allowed to continue in an open-label fashion to receive high-dose PXT3003 (receiving twice the low-dose for each administration (i.e. 10 mL). The objective is to mainly assess the safety and tolerability in the aforementioned patient population.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PXT3003 dose 1 (Active Comparator): Period 1, PXT3003 : Liquid oral solution (0.6 mg/mL baclofen, 0.07 mg/mL naltrexone HCl and 210 mg/mL D-sorbitol), 5 mL bid (taken morning and evening with food) for 9 consecutive months
  Interventions: Drug: PXT3003
- PXT3003 dose 2 (Active Comparator): Period 1, PXT3003: Liquid oral solution (1.2 mg/mL baclofen, 0.14 mg/mL naltrexone HCl and 420 mg/mL D-sorbitol), 5 mL bid (taken morning and evening with food) for 9 consecutive months
  Period 2, PXT3003: Liquid oral solution (0.6 mg/mL baclofen, 0.07 mg/mL naltrexone HCl and 210 mg/mL D-sorbitol), 10 mL bid (taken morning and evening with food)
  Interventions: Drug: PXT3003

INTERVENTIONS:
Drug: PXT3003 — Liquid oral solution, twice 5 mL (Dose 1) bid

SUMMARY:
All randomised patients with Charcot-Marie-Tooth Type 1A (CMT1A) who completed the primary study CLN-PXT3003-02, i.e. treatment with PXT3003 or placebo, are eligible to continue in the extension study CLN-PXT3003-03.

Period 1: Patients randomised to PXT3003 dose 1 or placebo in the primary study (CLN-PXT3003-02) continued in the extension study on PXT3003 dose 1 (5 mL). Patients randomised to PXT3003 dose 2 (5 mL) in the primary study (CLN-PXT3003-02) continued in the extension study on PXT3003 dose 2 or PXT3003 twice dose 1 (2x5 mL).

Period 2: All patients continue on twice dose 1 (2X5mL).

DETAILED DESCRIPTION:
PXT3003 is a rational design, fixed combination of low-dose (RS) baclofen, naltrexone hydrochloride and D-sorbitol. The use of PXT3003 in a multicenter, randomised, placebo controlled phase II study (CLN-PXT3003-01) was well-tolerated and safe in patients with CMT1A for the three dose-levels investigated (Attarian et al., 2014). The intermediate and high dose of PXT3003 demonstrated an improvement of disability in this patient population.

Subsequently a multicenter, randomised, placebo controlled phase III study (CLN-PXT3003-02) to assess the efficacy and safety of PXT3003 in the treatment of patients with CMT1A was initiated in December 2015. In March 2017 the first patients completed the 15-month treatment with PXT3003 and rolled over into the extension study CLN-PXT3003-03.

During Period 1 (9 months), patients that were randomised to PXT3003 dose 1 or placebo in the primary study (CLN-PXT3003-02) continued in the extension study on PXT3003 dose 1 (5 mL). Patients randomised to PXT3003 dose 2 (5 mL) in the primary study (CLN-PXT3003-02) continued in the extension study on on PXT3003 dose 2 or PXT3003 twice dose 1 (2x5 mL). During Period 2, all patients continue on twice dose 1 (2X5mL).

ELIGIBILITY:
Inclusion Criteria after September 18th 2017:

* Patients previously randomized to study CLN-PXT3003-02 under placebo and dose 1 and having completed 15 months of double-blind treatment in that study, including all procedures required at the Study Termination visit (V6) or
* Patients previously randomized to the initial study CLN-PXT3003-02 under dose 2, prematurely discontinued following sponsor decision, and having performed all procedures required at the Study Termination visit (V6)
* Patients whose V6 was performed within 4 weeks before entering the extension study or if not done must have a new baseline visit (VB)
* Female patients must agree to continue using an approved method of birth control throughout the extension study
* Patients must sign a written informed consent, specific to the extension study, in order to participate in this study. In case of minor children aged 16 to 18 years, both parent' and children's consents should be collected

Inclusion Criteria until September 18th 2017:

* Patients must have completed 15 months of double-blind treatment in the primary study CLN-PXT3003-02, including all procedures required at the Study Termination visit (V6)
* Female patients must agree to continue using an approved method of birth control throughout the extension study
* Patients must sign a written informed consent, specific to the extension study, in order to participate in this study. In case of minor children aged 16 to 18 years, both parent' and children's consents should be collected

Exclusion Criteria:

* Any clinically significant change in health status that, in the opinion of the Investigator, would prevent the subject from participating in this study or successfully completing this study
* Any unauthorized concomitant treatments, as study CLN-PXT3003-02 (e.g. including but not limited to baclofen, naltrexone,sorbitol (pharmaceutical form), opioids, levothyroxin, and potentially neurotoxic drugs such as amiodarone, chloroquine, cancer drugs susceptible to induce peripheral neuropathy)

Ages: 17 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) related to PXT3003 during the follow-up in patients with CMT1A | 9 or 24 months
  Incidence of treatment-emergent adverse events (TEAEs) related to PXT3003 during the follow-up in patients with CMT1A

SECONDARY OUTCOMES:
Incidence of all TEAEs and their evaluation of type/nature, severity/intensity, seriousness, duration, relationship to study drug, and outcome | 9 or 24 months
  Incidence of all TEAEs and their evaluation of type/nature, severity/intensity, seriousness, duration, relationship to study drug, and outcome
Incidence of adverse events leading to withdrawal of study drug | 9 or 24 months
  Incidence of adverse events leading to withdrawal of study drug
Overall Neuropathy Limitation Scale (ONLS) score, and its arm and leg sub-items | 9 or 24 months
  Overall Neuropathy Limitation Scale (ONLS) score, and its arm and leg sub-items
Charcot-Marie-Tooth Neuropathy Score - version 2 (CMTNS-V2), and its sub-items | 9 or 24 months
  Charcot-Marie-Tooth Neuropathy Score - version 2 (CMTNS-V2), and its sub-items
Nine-hole Peg Test (9-HPT) | 9 or 24 months
  Nine-hole Peg Test (9-HPT)
Quantified Muscular Testing (QMT) by hand grip and foot dorsiflexion dynamometry (mean of both sides) | 9 or 24 months
  Quantified Muscular Testing (QMT) by hand grip and foot dorsiflexion dynamometry (mean of both sides)
Time to walk 10 meters | 9 or 24 months
  Time to walk 10 meters
Compound Muscle Action Potential (CMAP) on ulnar nerve | 9 or 24 months
  Compound Muscle Action Potential (CMAP) on ulnar nerve
Sensory Nerve Action Potential (SNAP) on radial nerve | 9 or 24 months
  Sensory Nerve Action Potential (SNAP) on radial nerve
Nerve conduction velocity (NCV) | 9 or 24 months
  Nerve conduction velocity (NCV)
Quality of Life (EQ-5D) | 9 or 24 months
  Quality of Life (EQ-5D)
Visual analog scale on self-assessment of individualized main impairment in daily activities (defined at baseline with the patient) | 9 or 24 months
  Visual analog scale on self-assessment of individualized main impairment in daily activities (defined at baseline with the patient)

OTHER OUTCOMES:
Through plasma concentration of PXT3003 | at month 6 and 9
  Measurement of baclofen, naltrexone and 6-beta-naltrexone plasma concentration at the through
Peak plasma concentration of PXT3003 | at month 6 and 9
  Measurement of baclofen, naltrexone and 6-beta-naltrexone plasma concentration at the through

CONTACTS AND LOCATIONS:
Overall Officials: Shahram Attarian, MD, Principal Investigator — CHU la Timone, Marseille, France; Teresa Sevilla, MD, Principal Investigator — Hospital Universitario i Politécnico La F, Valencia, Spain; Marianne de Visser, MD, Principal Investigator — Academic Medical Center, Amsterdam, Netherlands; Mark Roberts, MD, Principal Investigator — Selor Royal NHS Foundation Trust, Manchester, UK; Florian Thomas, MD PhD, Principal Investigator — Seton Hall-Hackensack-Meridian School of Medicine, Hackensack, USA
Locations (23):
- United States (9):
  - Department of Neurology, Cedars-Sinai Medical Center, Los Angeles, California
  - Department of Neurology, McKnight Brain Institute, Gainesville, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Department of Neurology, University of Minnesota, Minneapolis, Minnesota
  - Department of Neurology and Psichiatry, Saint Louis University, St Louis, Missouri
  - Peripheral Neuropathy Center, Neurological Institue Building, Columbia University Medical Center, New York, New York
  - Saint Luke's Rehabilitation Institute, Spokane, Washington
- Departement of Neurology, UZ Leuven, Leuven, Belgium
- University Hospital of Quebec, Québec, Quebec, Canada
- France (6):
  - Cntre de Reference des Maladies Neuromusculaires, Hopital Swynghedauwl, CHU Lille, Lille
  - Centre de Reference des Neuropathies Peripheriques Rare, Hopital Dupuytren, CHU Limoges, Limoges
  - Service de Neurologie et du Sommeil, CHU Lyon Sud, Lyon
  - Centre de Reference des Maladie Neuromusculaires, CHU la Timone, Marseille
  - Centre de Reference des Maladie Neuromusculaires, Hotel Dieu, CHU de Nantes, Nantes
  - Service de Neurologie, Hopital Kremlin Bicetre, Paris
- Departement of Neurology, Academic Medical Center, Amsterdam, Netherlands
- Spain (4):
  - Department of neurology, Hospital Univesitario de Bellvitge, Barcelona
  - Servicio de Neurologia, Hospital Universitario La Paz, Madrid
  - Centro de Diagnostico y Tratamiento, Hospital Universitario Virgen del Rocio, Seville
  - Servicio de Neurologia, Hospital Universitario i Politécnic La Fe, Valencia
- Department of Neurology, Salford Royal NHS Foundation Trust, Salford, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No